CLINICAL TRIAL: NCT00166686
Title: Clonidine for the Treatment of Neurocognitive Sequelae Following Cancer Treatment in Children
Brief Title: Clonidine for Neurocognitive Sequelae
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PPRU 10706
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Treatment-Related Cancer
Keywords: Cancer; Clonidine; Neurocognitive sequelae
MeSH Terms: conditions — Neoplasms, Second Primary; Neoplasms | interventions — Clonidine

INTERVENTIONS:
Drug: Clonidine

SUMMARY:
The goals of the study are to determine the efficacy of clonidine in the treatment of children with neurocognitive sequelae following the therapy of long term malignancies. In addition, the study hopes to determine the long-term effect of clonidine on children's academic and psychosocial function.

DETAILED DESCRIPTION:
The long term prognosis for many children diagnosed with brain tumors and other malignancies has improved dramatically over the last decades and is expected to continue to rise as a result of improved treatment. The increased survival in pediatric oncology, however, has been associated with an increased recognition of neurobehavioral sequelae of cancer and its treatment. Current understanding of the incidence, pathogenesis, and natural history of these neurobehavioral abnormalities is limited and considerable individual variation in the presence and severity of these complications has been noted. Central nervous system (CNS) abnormalities associated with childhood cancer and its treatment have been demonstrated on at least three levels which may be interrelated: neurobehavioral abnormalities, brain imaging abnormalities, and neurotransmitter abnormalities.

Patients will be randomized to either clonidine or placebo. Study medication will be administered in a double blind fashion beginning with a four-week dose titration period followed by a four-week maintenance period. Total duration of dosing is 18 weeks. Patients who derive a benefit from clonidine administration may continue for an additional 30 weeks of therapy. PK samples will be collected at weeks 9 and 18.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a prior diagnosis of a pediatric malignancy (brain tumors, solid tumors, leukemia/lymphoma) who are in remission, and are > 3 years from initial diagnosis. Patients must have completed therapy a minimum of 6 months prior to study entry.
* Patients must have English as their primary language
* Patients must be >3 and less than or equal to 16 at the time of study enrollment
* Patients must fulfill the operational criteria for neurocognitive deficit and have an IQ > 50.
* Patients must be currently enrolled in a school or a learning environment where an adult familiar with the child's academic performance can provide ratings of that performance over the time of the trial.
* Patients must have wbc, hemoglobin and platelet parameters which fall within the norms for the patient's age.
* Patients must have adequate hepatic function (bilirubin less than or equal to 1.5 mg/dl and SGPT < 5x normal) and renal function (normal Cr for age/GFR greater than or equal to 70 ml/min/1.73m2)
* Patients must be able to swallow gel caps.
* Signed informed consent must be obtained according to institutional guidelines. When appropriate the patient will be included in all discussion in order to obtain verbal assent.
* Protocol and informed consent must be approved by the local IRB prior to any patient registration and reapproved every 12 months.

Exclusion Criteria:

* Patients who have evidence of a significant neurological abnormality prior to their cancer diagnosis that would affect neuro-behavioral development (such as genetic: Fragile X, Downs syndrome, or acquired disorders: closed head injury)
* Patients with a prior (pre-cancer) diagnosis of attention deficit hyperactivity disorder or major depression
* Patients who have a medical condition which would preclude the use of clonidine (medicated for hypertension, cardiac conduction disturbances, cerebrovascular disease, or chronic renal failure)
* Patients must not have received psychotropic medication (SSRIs, methylphenidate), anxiolytics, or hypnotics within 2 weeks of study entry.
* Patients who are receiving concurrent scheduled barbiturates or sedating drugs.
* Currently (within 6 months) known to abuse drugs or to be dependent on any drug including alcohol or with a positive urine drug screen.
* Women of childbearing age must not be pregnant or lactating. This group is excluded because of teratogenic potential of this agent demonstrated in rat and rabbit models.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States